CLINICAL TRIAL: NCT04728334
Title: A Multicenter, Phase 1, Dose Escalation and Dose Expansion Study to Evaluate the Safety, Pharmacokinetics, and Antitumor Activity of AK117 in Subjects With Advanced Solid Tumors or Lymphomas
Brief Title: A Phase 1 Dose Escalation and Expansion Study of AK117
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Akeso (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AK117-102
Record Dates: First submitted 2021-01-24; First posted 2021-01-28 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Neoplasms Malignant
Keywords: Antineoplastic Agents; Immunological
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AK117 monotherapy (Experimental): AK117 monotherapy intravenous (IV) infusion - Weekly doses
  Interventions: Drug: AK117

INTERVENTIONS:
Drug: AK117 — An intravenous (IV) infusion of AK117 as monotherapy. All subjects will receive 4 weekly infusions (Days 1, 8, 15, and 22) of AK117 in each 28-day treatment cycle until unacceptable toxicity, documentation of confirmed progressive disease (PD), or subject withdrawal

SUMMARY:
This is a multicenter, open label, single arm, Phase 1，dose escalation and dose expansion study designed to evaluate the safety, tolerability, pharmacodynamics, PK, immunogenicity, and preliminary antitumor activity of AK117 administered intravenously to adult subjects with relapsed/refractory advanced or metastatic solid tumors or lymphomas.

DETAILED DESCRIPTION:
The study comprises a dose escalation phase and a dose expansion phase. The phases will be conducted sequentially. Approximately 162 subjects will be enrolled in this study.

ELIGIBILITY:
Inclusion Criteria:

* All Subjects

  1. Able to provide written and signed informed consent and any locally required authorization obtained from the subject/legal representative, which must be obtained prior to performing any protocol related procedures.
  2. Men or women aged ≥18 years and ≤75 at the time of study entry.
  3. Eastern Cooperative Oncology Group (ECOG) performance status (PS) score of 0 or 1.
  4. Life expectancy ≥12 weeks.
  5. Willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures as specified in the protocol.
  6. Subjects must provide the tumor tissue samples after the diagnosis of solid tumor or lymphoma.
  7. Adequate organ function.
  8. Subjects with Solid Tumors：Subjects must have a histologically or cytologically confirmed advanced solid tumor that is refractory or relapsed to the current standard therapies, or for which no effective standard therapy is available. Subject must have at least 1 measurable lesion according to RECIST v1.1.
  9. Subjects with Lymphomas：Subjects must have histologically confirmed non-Hodgkin lymphoma(NHL), which may include transformed lymphoma, relapsed or refractory to autologous hematopoietic stem cell transplantation, or at least 2 lines of prior chemotherapy. Subjects must have disease that is measurable or assessable for response as per Lugano Classification 2014.

Exclusion Criteria:

* All Subjects

  1. Concurrent enrollment in another clinical study, unless it is an observational clinical study or the follow up period of an interventional study.
  2. Prior malignancy active within the previous 3 years except for the tumor for which a subject is enrolled in the study, and locally curable cancers that have been apparently cured.
  3. Receipt: The last cycle of anticancer therapy within 3 weeks prior to the first dose of investigational product; Anticancer small molecule targeted agent, palliative local treatment for non-target lesions, non-specific immunomodulatory therapy within 2 weeks prior to the first dose of investigational product; Chinese medicines with anti-tumor indications within 1 week prior to the first dose of investigational product; Any major surgery within 4 weeks; RBC infusion within 3 months.
  4. Metastasis or infiltration of brainstem and meninges;Metastasis or compression of the spinal cord; Active brain/central nervous system (CNS) metastases.
  5. Subjects with clinical symptoms or repeated drainage of pleural effusion, pericardial effusion or ascites.
  6. Cancer invasion of important surrounding organs or risk of esophageal tracheal fistula or esophageal pleural fistula.
  7. Known history of testing positive for human immunodeficiency virus (HIV) or known active acquired immunodeficiency syndrome.
  8. Known active hepatitis B or C infections (known positive HBsAg result or positive HCV antibody with detectable HCV ribonucleic acid [RNA] results).
  9. Active or prior documented autoimmune disease that may relapse.
  10. History of interstitial lung disease or noninfectious pneumonitis, except for those induced by radiation therapies.
  11. History of hemolytic anemia of any cause within 3 months prior to the first dose of investigational product.
  12. History of defects in RBC production, or hemoglobin production or metabolism.History of hemophagocytic lymphohistiocytosis.
  13. Previous or current gastrointestinal perforation, surgical incision, wound healing complications and bleeding events.
  14. Patients with clinically significant cardio-cerebrovascular disease.
  15. Unresolved toxicities from prior anticancer therapy, defined as having not resolved to NCI CTCAE v5.0 Grade 0 or 1, or to levels dictated in the eligibility criteria with the exception of toxicities not considered a safety risk.
  16. Subjects with a condition requiring systemic treatment with either corticosteroids or other immunosuppressive medications within 14 days prior to the first dose of investigational product.
  17. Subjects with prior use of anti-PD-1, anti-PD-L1, anti-CTLA-4, or any other immuno-oncology agents, receipt of the following treatments or procedures: Use of immunotherapy or IO drug within 21 days prior to the first dose; Subjects had an irAE that resulted in permanent discontinuation of previous immunotherapy; Subjects had a history of grade 3 or higher irAE or cardiac, neurological, or ocular irAE of any grade at the time of prior immunotherapy; Prior to screening in this study, all AEs at the time of previous immunotherapy had not been completely remission or remission to grade 1; Subjects need to use other immunosuppressants other than glucocorticoids systematically to treat irAE.
  18. History of severe hypersensitivity reactions to other mAbs.
  19. History of organ transplantation.
  20. Known allergy or reaction to any component of the investigational product formulation.
  21. Receipt any anticancer therapy targeting the CD47/SIRPα signaling axis.
  22. Known history of mental illness, alcohol or drug abuse.
  23. Existing uncontrolled comorbiditions; Or a mental illness/social condition that may limit the subject's compliance with study requirements or affect the subject's ability to provide written informed consent.
  24. Other exclusion criteria for subjects with lymphoma:History of HTLV-1 infection.Subjects with primary or secondary central nervous system lymphoma. Subjects with history of allogeneic hematopoietic stem cell transplantation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2021-03-23 (Actual); Primary Completion 2022-01-25 (Actual); Study Completion 2023-05-12 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events (AEs) | From the time of informed consent signed through 30 days after the last dose of AK117
  An AE is defined as any untoward medical occurrence in a participant administered a pharmaceutical product temporally associated with the use of study treatment, whether or not considered related to the study treatment.
Number of participants with a Dose Limiting Toxicity (DLT) | During the first 21 days
  DLTs will be assessed during the first 21 days of treatment for dose-escalation phase and are defined as toxicities that meet pre-defined severity criteria, and assessed as having a suspected relationship to study drug, and unrelated to disease, disease progression, inter-current illness, or concomitant medications .

SECONDARY OUTCOMES:
Objective response rate (ORR) | Up to 2 years
  ORR defined as the proportion of subjects who achieves a best overall response of CR or PR, assessed by Investigator per RECIST Version 1.1 for solid tumor or the Lugano 2014 Classification for lymphoma
Disease control rate (DCR) | Up to 2 years
  The DCR is defined as the proportion of subjects with CR, PR, or SD .
Maximum observed concentration (Cmax) of AK117 | From first dose of AK117 through to 30 days after last dose of AK117
  The endpoints for assessment of PK of AK104 include serum concentrations of AK117 at different timepoints after AK117 administration.
Minimum observed concentration (Cmin) of AK117 at steady state | From first dose of AK117 through to 30 days after last dose of AK117
  The endpoints for assessment of PK of AK104 include serum concentrations of AK117 at different timepoints after AK117 administration.
Number of subjects who develop detectable anti-drug antibodies (ADAs) | From first dose of AK117 through to 30 days after last dose of AK117
  The immunogenicity of AK117 will be assessed by summarizing the number of subjects who develop detectable antidrug antibodies (ADAs).

CONTACTS AND LOCATIONS:
Overall Officials: Jiong Wu, MD, Principal Investigator — Fudan University
Locations (1):
- FuDan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No